CLINICAL TRIAL: NCT01556919
Title: Development of an Esophageal Monitoring Device for the Assessment of Esophageal Epithelium Integrity With Mucosal Impedance
Brief Title: Esophageal Monitoring Device for Assessing Mucosal Impedance
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Medical Director, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 120126
Record Dates: First submitted 2012-03-12; First posted 2012-03-19 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: GERD; Esophagitis
Keywords: GERD; Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mucosal Impedance Probe
  Interventions: Procedure: Standard of care endoscopy

INTERVENTIONS:
Procedure: Standard of care endoscopy — standard of care endoscopy

SUMMARY:
The investigators are looking at a novel approach to measuring gastroesophageal reflux disease (GERD) damage and reducing the need for costly and less optimal testing presently used for diagnostic and treatment purposes. The investigators will be using three custom mucosal impedance (MI) catheters, each designed to measure at slightly different spacing on the esophagus.

DETAILED DESCRIPTION:
During routine esophagogastroduodenoscopy (EGD), consented study participants will have a series of three (3) custom mucosal impedance (MI) catheters with an axial array of sensors positioned along the mucosal wall to directly measure mucosal impedance at various intervals. Each catheter will be manually guided by the physician through the working channel of the endoscope until the sensored tip is visible through the scope camera. The physician will place the sensored rings directly on the mucosa along the lumen. To obtain evaluable data, the sensors must remain in contact with the mucosa at each point for 5 seconds after a stable impedance reading has been captured. This process will be repeated for each of the three prototype catheters in each consented patient in order to determine the optimal catheter/sensor design. The catheters will be attached to a channeled feed that will record measurements on a dedicated computer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing standard of care EGD with or without BRAVO placement;
* Have GERD symptoms and/or have endoscopic esophagitis

Exclusion Criteria:

* Use of acid suppressive therapy within last 10 days;
* Known history of Barrett's esophagus, gastric surgery, alcoholism, significant motility condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for an esophagogastroduodenoscoy (EGD) for one of the following reasons: diagnosed with Gastroesophegeal reflux disease (GERD); have a normal esophageal mucosa but an abnormal pH testing (acid measurement); or a normal esophagus and normal pH testing
Sampling Method: Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2012-03; Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Mucosal Impedance Values | Values will be obtained at conclusion of EGD, an expected average of 5 minutes
  Consented study participants will have a series of three (3) custom mucosal impedance (MI) catheters with an axial array of sensors positioned along the mucosal wall to directly measure mucosal impedance at various intervals. The catheters will be attached to a channeled feed that will record measurements on a dedicated computer.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center Endoscopy Laboratory, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Ates F, Yuksel ES, Higginbotham T, Slaughter JC, Mabary J, Kavitt RT, Garrett CG, Francis D, Vaezi MF. Mucosal impedance discriminates GERD from non-GERD conditions. Gastroenterology. 2015 Feb;148(2):334-43. doi: 10.1053/j.gastro.2014.10.010. Epub 2014 Oct 16. PMID 25448923